CLINICAL TRIAL: NCT04409392
Title: Staphylococcus Lugdunensis Prosthetic Joint Infection: a Retrospective Cohort Study
Brief Title: Staphylococcus Lugdunensis Prosthetic Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20-202
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-11

CONDITIONS: Staphylococcal Infections; Prosthetic Joint Infection
Keywords: Staphylococcus lugdunensis; Prosthetic Joint Infection; biofilm
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prothestic joint infection due to Staphylococcus lugdunensis: Patients having had a prosthetic joint infection with Staphylococcus lugdunensis
  Interventions: Other: Prothestic joint infection due to Staphylococcus lugdunensis

INTERVENTIONS:
Other: Prothestic joint infection due to Staphylococcus lugdunensis — description of prosthetic joint infection with Staphylococcus lugdunensis

SUMMARY:
Staphylococcus lugdunensis is a coagulase-negative staphylococcus belonging to the human commensal cutaneous flora, and has been little studied in the field of prosthetic joint infections. However, it shares many virulence traits with Staphylococcus aureus, including many adhesins and its ability to form biofilm, and the few series of cases reports a significant failure rate.

ELIGIBILITY:
Inclusion Criteria:

* infection of joint prosthesis (whatever its type) with Staphylococcus lugdunensis defined by the positivity of at least 2 gold-standard samples (joint puncture, intraoperative samples) with S. lugdunensis; OR
* a single positive gold-standard sample or positive blood cultures AND formal clinical, radiological, biological and / or pathological arguments in favor of an infection of joint prosthesis AND absence of other pathogenic agent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having had IPA due to Staphylococcus lugdunensis
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of PJI infection with Staphylococcus lugdunensis | between 2010 and 2020
  proportion of patients having PJI infection with Staphylococcus lugdunensis, alone or with other bacteria
Description of PJI infection with Staphylococcus lugdunensis : type | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  type of PJI : knee or hip prosthesis
Description of PJI infection with Staphylococcus lugdunensis : evolution | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  evolution of PJI :evolution between prosthesis placement and the onset of symptoms, gateway to infection
Description of patients with PJI infection due to Staphylococcus lugdunensis | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  type of patients: age, CMI
Description of patients with PJI infection due to Staphylococcus lugdunensis : follow up | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  duration of the follow up of patients
Description of patients with PJI infection due to Staphylococcus lugdunensis : medical treatment | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  description and duration of antibiotics
Description of patients with PJI infection due to Staphylococcus lugdunensis : surgical treatment | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  description of surgery performed : DAIR, one-step exchange, two-step exchange
rate of treatment failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr